CLINICAL TRIAL: NCT03631147
Title: The Effect of Rifaximin on Portal Vein Thrombosis in Cirrhotic Patients
Brief Title: The Effect of Rifaximin on Portal Vein Thrombosis
Acronym: ERPVT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Shiyao Chen, Professor, Shanghai Zhongshan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CSY-RFXM-PVT
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Cirrhosis; Portal Vein Thrombosis
MeSH Terms: conditions — Fibrosis | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rifaximin treatment group (Experimental): Rifaximin 400mg bid for 8 weeks
  Interventions: Drug: Rifaximin
- The control group (No Intervention)

INTERVENTIONS:
Drug: Rifaximin — 400mg bid for 8 weeks
  Other Names: XIFAXAN
  Arms: Rifaximin treatment group

SUMMARY:
The aim of this study is to evaluate the efficacy of rifaximin in the treatment of portal vein thrombosis in cirrhotic patients

DETAILED DESCRIPTION:
Portal vein thrombosis is not an uncommon complication in cirrhotic portal hypertension, which lead to a poor prognosis in endoscopic management of variceal bleeding. Evidence indicated that enoxaparin prevented PVT and liver decompensation via decreased rates of bacterial infections and lowered the potent inflammatory mediators such as interleukin-6. Rifaximin is a broad-spectrum antibiotic that exerts endotoxin-lowering and anti-inflammatory effects.

ELIGIBILITY:
Inclusion Criteria:

* 18 y.o. ≤age≤75 y.o
* Cirrhotic patients had CTA confirmed portal vein trombosis
* D-dimer no more than five times the normal upper limit

Exclusion Criteria:

* age <18 y.o. or age > 75 y.o.
* had portal cavernoma
* received anticoagulation treatment in the past 6 months
* splenectomy
* Known infection after endoscopic treatment (Fever, microbial cultures positive, et al.)
* Massive ascites or combined with other high risk factor that require prophylaxis use of antibiotics.
* Acute variceal bleeding within 5 days.
* Use of other antibiotics in the past 2 weeks
* Acute portal vein thrombosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2018-09-03 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes of portal vein thrombosis | 8 weeks
  The changes of portal vein thrombosis in 8 weeks (include main portal vein, left and/or right portal vein, superior mesenteric vein, et al)

SECONDARY OUTCOMES:
Changes of portal vein thrombosis | 6 months
  The changes of portal vein thrombosis in 8 weeks (include main portal vein, left and/or right portal vein, superior mesenteric vein, et al)
All clinical events | 8 weeks
  All clinical events were defined as occurrence rebreeding, ascitic fluid infection, hepatorenal syndrome, hepatopulmonary syndrome, portal vein thrombosis, or death
All clinical events | 6 months
  All clinical events were defined as occurrence rebreeding, ascitic fluid infection, hepatorenal syndrome, hepatopulmonary syndrome, portal vein thrombosis, or death

CONTACTS AND LOCATIONS:
Locations (1):
- 180 Fenglin Road, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qi X, Han G, Fan D. Management of portal vein thrombosis in liver cirrhosis. Nat Rev Gastroenterol Hepatol. 2014 Jul;11(7):435-46. doi: 10.1038/nrgastro.2014.36. Epub 2014 Apr 1. PMID 24686266
- [Background] Mantaka A, Augoustaki A, Kouroumalis EA, Samonakis DN. Portal vein thrombosis in cirrhosis: diagnosis, natural history, and therapeutic challenges. Ann Gastroenterol. 2018 May-Jun;31(3):315-329. doi: 10.20524/aog.2018.0245. Epub 2018 Mar 3. PMID 29720857
- [Background] Qi X, Bai M, Yang Z, Yuan S, Zhang C, Han G, Fan D. Occlusive portal vein thrombosis as a new marker of decompensated cirrhosis. Med Hypotheses. 2011 Apr;76(4):522-6. doi: 10.1016/j.mehy.2010.12.007. Epub 2011 Jan 8. PMID 21216538
- [Background] D'Amico G, De Franchis R; Cooperative Study Group. Upper digestive bleeding in cirrhosis. Post-therapeutic outcome and prognostic indicators. Hepatology. 2003 Sep;38(3):599-612. doi: 10.1053/jhep.2003.50385. PMID 12939586
- [Background] Cruz-Ramon V, Chinchilla-Lopez P, Ramirez-Perez O, Aguilar-Olivos NE, Alva-Lopez LF, Fajardo-Ordonez E, Ponciano-Rodriguez G, Northup PG, Intagliata N, Caldwell SH, Qi X, Mendez-Sanchez N. Thrombosis of the Portal Venous System in Cirrhotic vs. Non-Cirrhotic Patients. Ann Hepatol. 2018 May-June;17(3):476-481. doi: 10.5604/01.3001.0011.7392. Epub 2018 Apr 9. PMID 29735798
- [Background] Kimer N, Pedersen JS, Tavenier J, Christensen JE, Busk TM, Hobolth L, Krag A, Al-Soud WA, Mortensen MS, Sorensen SJ, Moller S, Bendtsen F; members of the CoRif study group. Rifaximin has minor effects on bacterial composition, inflammation, and bacterial translocation in cirrhosis: A randomized trial. J Gastroenterol Hepatol. 2018 Jan;33(1):307-314. doi: 10.1111/jgh.13852. PMID 28671712
- [Background] Bajaj JS. Review article: potential mechanisms of action of rifaximin in the management of hepatic encephalopathy and other complications of cirrhosis. Aliment Pharmacol Ther. 2016 Jan;43 Suppl 1:11-26. doi: 10.1111/apt.13435. PMID 26618922